CLINICAL TRIAL: NCT04439513
Title: Randomized Comparison f Dual Artery Compression Versus Radial Artery-Only Hemostasis: Impact on Radial Artery Occlusion (EArly Discharge After Transradial Stenting of coronarY Arteries - EASY-RAO)
Brief Title: Dual Artery Compression vs. Radial Artery-Only Hemostasis: Impact on Radial Artery Occlusion (EASY-RAO)
Acronym: EASY-RAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olivier F. Bertrand (Other)
Responsible Party: Sponsor-Investigator, Olivier F. Bertrand, Director of the International Chair on Interventional Cardiology and Transradial Approach, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EASY-RAO; 2020-3400, 21885 (Other: IUCPQ)
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Radial Artery Injury
Keywords: RAO; Hemostasis; TRA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Artery Compression (Experimental): time to hemostasis and incidence of radial artery occlusion will be monitored while using a dual artery compression device (Terry-2-band) to achieve hemostasis.
  Interventions: Device: Hemostasis
- Radial Artery-Only (Active Comparator): time to hemostasis and incidence of radial artery occlusion will be monitored while using the device currently approved by the institution (Hemo-Stop) and following institutional protocols for hemostasis.
  Interventions: Device: Hemostasis

INTERVENTIONS:
Device: Hemostasis — Compression device to achieve hemostasis.

SUMMARY:
This study aims to demonstrate the superiority in clinical performances of a dual artery compression device (Terry-2 band) compared to a standard radial artery-only hemostasis device (HemoSTOP).

ELIGIBILITY:
Inclusion Criteria:

* any patients referred for diagnostic angiography and possible percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Patient unable to understand study design or objectives
* Unable to sign informed consent
* Patient taking warfarin or other anticoagulant therapy
* Chronic RAO on both sides precluding TRA
* Previous ipsilateral transradial approach
* Inability to comply with the study follow-up
* Presence of plethysmographic waveform with radial and ulnar occlusive compression
* Pre-existing local complication (i.e. hematoma, pseudo-aneurysm, ...) precluding access-site evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Rate of RAO after transradial approach (TRA) at hospital discharge | up to 24 hours
  To determine whether the use of a dual artery compression decreases the rate of radial artery occlusion after transradial catheterization.

SECONDARY OUTCOMES:
Percentage of radial artery patent-hemostasis during hemostasis | throughout intervention, up to 180 minutes
  To determine the conservation of blood flow through the radial artery during compressive hemostasis
Patient comfort during hemostasis as assessed on a visual scale | throughout intervention, up to 30 days
  To evaluate the level of patient comfort in relation to the device used
Rates of complications such as repeat bleeding and hematoma (EASY Scale) | throughout intervention, up to 30 days
  To determine the incidence of complications in relation to the device used. Bleeding, spasm and presence of hematomas will be evaluated.
Nursing involvement in hemostasis management for sensitivity analysis on cost assessment | throughout intervention, up to 24 hours
  To determine the overall nursing involvement (time per nurse per patient) in hemostasis monitoring from end of procedure to patient discharge for a cost-benefit evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCPQ - Laval Hospital, Québec, Canada

IPD SHARING:
Plan to Share IPD: No